CLINICAL TRIAL: NCT01369498
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of GS-6624 in Adult Subjects With Primary, Post Polycythemia Vera or Post Essential Thrombocythemia Myelofibrosis
Brief Title: Efficacy and Safety of Simtuzumab in Adults With Primary, Post Polycythemia Vera or Post Essential Thrombocythemia Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB0024-102; NCT01242709 (obsolete NCT alias)
Record Dates: First submitted 2011-06-06; First posted 2011-06-09 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Myelofibrosis
Keywords: Hematology; Myelofibrosis; Thrombocythemia Myelofibrosis; Bone Marrow Diseases; Hematologic Diseases; Blood Diseases; Leukemia; Blood Disorders
MeSH Terms: conditions — Primary Myelofibrosis; Bone Marrow Diseases; Hematologic Diseases; Leukemia | interventions — simtuzumab; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Simtuzumab 200 mg (Experimental): Participants in Stage 1 of study will receive simtuzumab 200 mg for up to 24 weeks. Treatment could be continued if there is evidence of clinical benefit as judged by the treating physician.
  Interventions: Drug: Simtuzumab
- Simtuzumab 700 mg (Experimental): Participants in Stage 1 of study will receive simtuzumab 700 mg for up to 24 weeks. Treatment could be continued if there is evidence of clinical benefit as judged by the treating physician.
  Interventions: Drug: Simtuzumab
- Simtuzumab 200 mg+Ruxolitinib (Experimental): In Stage 2, participants on stable doses of ruxolitinib will receive simtuzumab 200 mg for at least 24 weeks. Treatment could be continued if there is evidence of clinical benefit as judged by the treating physician.
  Interventions: Drug: Simtuzumab; Drug: Ruxolitinib
- Simtuzumab 700 mg+Ruxolitinib (Experimental): In Stage 2, participants on stable doses of ruxolitinib will receive simtuzumab 700 mg for at least 24 weeks. Treatment could be continued if there is evidence of clinical benefit as judged by the treating physician.
  Interventions: Drug: Simtuzumab; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Simtuzumab — Simtuzumab administered intravenously over approximately 30 minutes every 2 weeks
  Other Names: GS-6624; AB0024
Drug: Ruxolitinib — In Stage 2, participants will be on a stable dose of ruxolitinib
  Arms: Simtuzumab 200 mg+Ruxolitinib; Simtuzumab 700 mg+Ruxolitinib

SUMMARY:
This study is to evaluate the efficacy and safety of simtuzumab (GS-6624) on bone marrow fibrosis either alone or in combination with ruxolitinib in participants with primary myelofibrosis (PMF) and post polycythemia vera or post essential thrombocythemia myelofibrosis (ET/PV MF).

The study is designed as a two-stage trial. In the stage 1, participants will be randomized into two cohorts to receive either 200 or 700 mg of study drug. In the stage 2, participants on ruxolitinib will be randomized to receive either 200 or 700 mg of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with PMF or post ET/PV MF with intermediate-1, intermediate-2 or high risk disease according to the international working group (IWG) prognostic scoring system, or if with low risk disease then with symptomatic splenomegaly that is ≥ 10 cm below left costal margin by physical exam.
* Must have adequate organ function as demonstrated by the following:
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 2.5x upper limit of normal (ULN), or ≤ 4x ULN (if upon judgment of the treating physician, it is believed to be due to extramedullary hematopoiesis [EMH] related to MF);
* Direct bilirubin ≤ 1.5 x ULN; or ≤ 2x ULN (if upon judgment of the treating physician, it is believed to be due to extramedullary hematopoiesis [EMH] related to MF);
* Serum creatinine ≤ 2.5 mg/dL.
* In Stage 2, participants must be on ruxolitinib for at least 8 weeks and on a stable dose for at least 4 weeks.
* Eastern cooperative oncology group (ECOG) performance status (PS) ≤ 2
* Treatment-related toxicities from prior therapies must have resolved to Grade ≤ 1
* Women of childbearing potential and men must agree to using one medically approved (ie, mechanical or pharmacological) contraceptive measure and have their partners agree to an additional barrier method of contraception for the duration of the study and for 90 days after the last administration of study drug. Definition of female of child bearing potential and a list of acceptable contraceptive methods for this study applies per protocol.

Exclusion Criteria:

* Any serious medical condition or psychiatric illness that would prevent, (as judged by the treating physician) the participant from signing the informed consent form or any condition, including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Pregnant or lactating.
* Known history of human immunodeficiency virus (HIV), hepatitis C, or hepatitis B.
* History or presence of any form of cancer within the 3 years prior to enrollment, with the exception of excised basal cell or squamous cell carcinoma of the skin, or cervical carcinoma in situ or breast carcinoma in situ that has been excised or resected completely and is without evidence of local recurrence or metastasis.
* Participation in an investigational drug or device trial within 2 weeks prior to study Day 1 or within 5 times the half-life of the investigational agent in the other clinical study, if known.
* Use of any cytotoxic chemotherapeutic agents (eg, hydroxyurea), corticosteroids (prednisone ≤ 10 mg/day or corticosteroid equivalent is allowed), or immune modulators (eg, thalidomide) within 2 weeks and interferon use within 4 weeks prior to study Day 1.
* Symptomatic congestive heart failure (New York Heart Association Classification > Class II), unstable angina, or unstable cardiac arrhythmia requiring medication.
* History of surgery within 2 weeks prior to enrollment or anticipated surgery during the study period.
* Any other condition that might reduce the chance of obtaining data required by the protocol or that might compromise the ability to give truly informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-06-30 (Actual); Primary Completion 2014-06-05 (Actual); Study Completion 2014-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (7):
- United States (7):
  - Mayo Clinic, Scottsdale, Arizona
  - Stanford University Medical center, Stanford, California
  - Washington University in St. Louis, St Louis, Missouri
  - Oncology Hematology Care Clinical Trials, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 30 June 2011. The last study visit occurred on 24 September 2014.
Pre-assignment Details: 62 participants were screened.
Groups:
- Stage 1: SIM 200 mg: Participants were administered simtuzumab (SIM) 200 mg intravenous (IV) infusion over 30 minutes once every 2 weeks for a total of 6 infusions per 12-week cycle for up to 94 weeks.
- Stage 1: SIM 700 mg: Participants were administered SIM 700 mg IV infusion over 30 minutes once every 2 weeks for a total of 6 infusions per 12-week cycle for up to 40 weeks.
- Stage 2: SIM 200 mg+Ruxolitinib: Participants on a stable dose of ruxolitinib were administered SIM 200 mg IV infusion over 30 minutes once every 2 weeks for up to 91 weeks.
- Stage 2: SIM 700 mg+Ruxolitinib: Participants on a stable dose of ruxolitinib were administered SIM 700 mg IV infusion over 30 minutes once every 2 weeks for up to 86 weeks.
Period: Overall Study
Arm/Group | Stage 1: SIM 200 mg | Stage 1: SIM 700 mg | Stage 2: SIM 200 mg+Ruxolitinib | Stage 2: SIM 700 mg+Ruxolitinib
Started | 12 | 12 | 15 | 15
Completed | 0 | 0 | 0 | 0
Not Completed | 12 | 12 | 15 | 15
Not completed — Lack of Efficacy | 9 | 9 | 1 | 3
Not completed — Adverse Event | 1 | 2 | 0 | 1
Not completed — Withdrawal of Consent | 0 | 1 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Investigator's Discretion | 1 | 0 | 1 | 3
Not completed — Unknown Reason | 1 | 0 | 11 | 6
Not completed — Disease Progression | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1: SIM 200 mg | Stage 1: SIM 700 mg | Stage 2: SIM 200 mg+Ruxolitinib | Stage 2: SIM 700 mg+Ruxolitinib | Total
Number analyzed (Participants) | 12 | 12 | 15 | 15 | 54
Age, Customized [Count of Participants; unit: Participants]
  Age: > 65 years | 9 | 8 | 12 | 9 | 38
  Age: ≤ 65 years | 3 | 4 | 3 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 9 | 4 | 23
  Male | 6 | 8 | 6 | 11 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 12 | 11 | 15 | 14 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 12 | 11 | 13 | 14 | 50
  Race: Black or African Heritage | 0 | 1 | 0 | 1 | 2
  Race: Other | 0 | 0 | 1 | 0 | 1
  Race: Asian | 0 | 0 | 1 | 0 | 1
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Race: Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0
Bone Marrow Fibrosis Score [Count of Participants; unit: Participants] — Population: The Per Protocol Analysis Set included participants who were randomized, received at least 1 dose of study drug, did not violate any major entry criteria and had at least 80% adherence with study drug. It is measured on a scale of 0-3 where 0 indicates normal marrow and 3 indicates fibrosis. For additional description, please see outcome measure 1.
  Participants
    number analyzed (Participants) | 11 | 12 | 15 | 15 | 53
    MF-0 | 0 | 0 | 0 | 0 | 0
    MF-1 | 2 | 1 | 1 | 3 | 7
    MF-2 | 4 | 2 | 6 | 5 | 17
    MF-3 | 5 | 8 | 8 | 7 | 28
    Missing | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Clinical Response as Defined by the Percentage of Participants With Reduction at Week 24 From Baseline in the Bone Marrow Fibrosis Score
Description: Overall response for the study drug is defined by the reduction in bone marrow fibrosis score which is on a scale of 0-3 where 0 indicates the scattered linear reticulin with no fiber intersections representing normal marrow and 3 indicates dense increase in reticulin fibrosis with fiber intersections, often with osteosclerosis. Reduction from baseline of score indicates improvement in clinical condition.
Time Frame: Baseline; Week 24
Population: The Per Protocol Analysis Set included participants who were randomized, received at least 1 dose of study drug, did not violate any major entry criteria, and had at least 80% adherence with study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: SIM 200 mg | Stage 1: SIM 700 mg | Stage 2: SIM 200 mg+Ruxolitinib | Stage 2: SIM 700 mg+Ruxolitinib
Number analyzed (Participants) | 11 | 12 | 15 | 15
percentage of participants | 0 [0.0 to 23.8] | 16.7 [3.0 to 43.8] | 6.7 [0.3 to 27.9] | 13.3 [2.4 to 36.3]

2. Secondary Outcome: Rate of Clinical Response as Defined by the Percentage of Participants With Improvement in Hemoglobin, Platelet, or Absolute Neutrophil Count (ANC)
Description: Overall response for the study drug was defined by the rate of clinical improvement in hemoglobin, platelet or ANC. Clinical improvement in hemoglobin was defined as a ≥ 2 g/dL increase from baseline in hemoglobin level and transfusion independent (absence of red blood cell (RBC) transfusions in prior 8 weeks and applicable only for participants with baseline hemoglobin level of < 10 g/dL); clinical improvement in platelets was defined as a ≥ 100% increase from baseline in platelet count and an absolute platelet count of ≥ 50 x 10^9/L (applicable only for participants with baseline platelet count < 50 x 10^9/L); clinical improvement in ANC is defined as a ≥ 100% increase from baseline in ANC and an ANC of ≥ 0.5 x 10^9/L (applicable only for participants with baseline ANC < 1 x 10^9/L).
Time Frame: Baseline; Weeks 12, 24 and any time post baseline (enrollment up to 94 weeks)
Population: Participants in Per Protocol Analysis Set with available data were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Stage 1: SIM 200 mg: Participants were administered SIM 200 mg IV infusion over 30 minutes once every 2 weeks for a total of 6 infusions per 12-week cycle for up to 94 weeks.
Arm/Group | Stage 1: SIM 200 mg | Stage 1: SIM 700 mg | Stage 2: SIM 200 mg+Ruxolitinib | Stage 2: SIM 700 mg+Ruxolitinib
Number analyzed (Participants) | 10 | 10 | 9 | 10
percentage of participants
  Week 12 | 0 [0.0 to 25.9] | 0 [0.0 to 25.9] | 0 [0.0 to 28.3] | 0 [0.0 to 25.9]
  Week 24 | 0 [0.0 to 25.9] | 0 [0.0 to 25.9] | 0 [0.0 to 28.3] | 0 [0.0 to 25.9]
  Any Time Post-Baseline | 0 [0.0 to 25.9] | 0 [0.0 to 25.9] | 11.1 [0.6 to 42.9] | 0 [0.0 to 25.9]

3. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: First dose date up to the last dose date (maximum: 94 weeks) plus 28 days
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1: SIM 200 mg | Stage 1: SIM 700 mg | Stage 2: SIM 200 mg+Ruxolitinib | Stage 2: SIM 700 mg+Ruxolitinib
Number analyzed (Participants) | 12 | 12 | 15 | 15
percentage of participants | 100 | 100 | 100 | 100

4. Secondary Outcome: Change From Baseline in Myelofibrosis Symptoms Assessment Score
Description: Myelofibrosis symptom assessment was performed using myeloproliferative neoplasm symptoms assessment form (MPN-SAF) which is a 27-item questionnaire to address symptom burden and quality of life. The form consists of 27 questions which are scored on a scale of 0-10 by participants based on how symptoms are affecting them, where 0 indicates less symptoms while 10 indicated more severe symptoms and greater inactivity. The MPN-SAF score was calculated at each visit for each participant as an average of the scales for each question and all answered questions. If the number of questions not answered at 1 visit was > 10, then the MPN-SAF score for that visit was taken as missing. A negative change from Baseline indicated improvement.
Time Frame: Baseline; Days 43 and 85 of Cycles 1-7 (cycle=12 weeks)
Population: Participants in the Per Protocol Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: SIM 200 mg | Stage 1: SIM 700 mg | Stage 2: SIM 200 mg+Ruxolitinib | Stage 2: SIM 700 mg+Ruxolitinib
Number analyzed (Participants) | 11 | 12 | 13 | 14
score on a scale
  Baseline | 2.5 (1.75) | 3.7 (1.86) | 3.2 (2.06) | 2.2 (1.34)
  Best Change from Baseline: number analyzed (Participants) | 9 | 11 | 13 | 13
  Best Change from Baseline | -0.9 (1.11) | -1.3 (1.60) | -1.1 (1.25) | -0.6 (0.98)
  Change from Baseline at Cycle 1 - Day 43: number analyzed (Participants) | 9 | 10 | 13 | 12
  Change from Baseline at Cycle 1 - Day 43 | -0.2 (0.58) | -1.0 (1.66) | -0.2 (0.81) | 0.2 (1.00)
  Change from Baseline at Cycle 1 - Day 85: number analyzed (Participants) | 9 | 10 | 12 | 11
  Change from Baseline at Cycle 1 - Day 85 | -0.3 (1.59) | -0.9 (1.67) | 0.5 (1.36) | 0.4 (0.74)
  Change from Baseline at Cycle 2 - Day 43: number analyzed (Participants) | 7 | 7 | 12 | 12
  Change from Baseline at Cycle 2 - Day 43 | -0.3 (0.99) | -1.0 (1.26) | -0.7 (1.30) | 0.4 (1.43)
  Change from Baseline at Cycle 2 - Day 85: number analyzed (Participants) | 7 | 6 | 11 | 10
  Change from Baseline at Cycle 2 - Day 85 | 0.3 (0.89) | -0.8 (1.44) | -0.5 (1.42) | 0.7 (1.61)
  Change from Baseline at Cycle 3 - Day 43: number analyzed (Participants) | 3 | 2 | 10 | 5
  Change from Baseline at Cycle 3 - Day 43 | 1.1 (2.81) | -1.2 (2.33) | -0.5 (1.16) | -0.3 (0.58)
  Change from Baseline at Cycle 3 - Day 85: number analyzed (Participants) | 2 | 2 | 8 | 5
  Change from Baseline at Cycle 3 - Day 85 | 0.1 (1.10) | 0.6 (1.55) | -0.5 (1.22) | -0.8 (0.39)
  Change from Baseline at Cycle 4 - Day 43: number analyzed (Participants) | 1 | 0 | 9 | 4
  Change from Baseline at Cycle 4 - Day 43 | 0 (NA) — Standard deviation was not calculated due to low number of participants |  | -0.4 (1.35) | -0.6 (1.29)
  Change from Baseline at Cycle 4 - Day 85: number analyzed (Participants) | 1 | 0 | 8 | 4
  Change from Baseline at Cycle 4 - Day 85 | 1.2 (NA) — Standard deviation was not calculated due to low number of participants |  | -0.8 (1.46) | -0.2 (0.68)
  Change from Baseline at Cycle 5 - Day 43: number analyzed (Participants) | 1 | 0 | 7 | 3
  Change from Baseline at Cycle 5 - Day 43 | 1.8 (NA) — Standard deviation was not calculated due to low number of participants |  | -0.6 (1.22) | -0.9 (0.53)
  Change from Baseline at Cycle 5 - Day 85: number analyzed (Participants) | 1 | 0 | 5 | 3
  Change from Baseline at Cycle 5 - Day 85 | 1.0 (NA) — Standard deviation was not calculated due to low number of participants |  | -1.2 (1.24) | -0.9 (0.91)
  Change from Baseline at Cycle 6 - Day 43: number analyzed (Participants) | 1 | 0 | 5 | 3
  Change from Baseline at Cycle 6 - Day 43 | 1.4 (NA) — Standard deviation was not calculated due to low number of participants |  | -0.4 (0.65) | -0.5 (0.32)
  Change from Baseline at Cycle 6 - Day 85: number analyzed (Participants) | 0 | 0 | 3 | 1
  Change from Baseline at Cycle 6 - Day 85 |  |  | -1.5 (0.84) | -0.9 (NA) — Standard deviation was not calculated due to low number of participants
  Change from Baseline at Cycle 7 - Day 43: number analyzed (Participants) | 0 | 0 | 1 | 1
  Change from Baseline at Cycle 7 - Day 43 |  |  | -1.4 (NA) — Standard deviation was not calculated due to low number of participants | -1.4 (NA) — Standard deviation was not calculated due to low number of participants
  Change from Baseline at Cycle 7 - Day 85: number analyzed (Participants) | 0 | 0 | 1 | 0
  Change from Baseline at Cycle 7 - Day 85 |  |  | -1.3 (NA) — Standard deviation was not calculated due to low number of participants |

5. Secondary Outcome: Change From Baseline in Cytokine Levels
Description: Biomarker samples were collected to evaluate the effects of SIM treatment on markers of serum and plasma cytokines.
Time Frame: Baseline; Week 24
Population: The cytokine analysis was not performed.
Arm/Group | Stage 1: SIM 200 mg | Stage 1: SIM 700 mg | Stage 2: SIM 200 mg+Ruxolitinib | Stage 2: SIM 700 mg+Ruxolitinib
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With Anti-Simtuzumab Antibody Formation
Description: Blood samples were collected for the presence of anti-SIM antibodies which was determined using a validated electro-chemiluminescent (ECL) assay screening test.
Time Frame: Baseline; Day 85 of Cycles 1 to 5 (cycle=12 weeks)
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Stage 1: SIM 200 mg | Stage 1: SIM 700 mg | Stage 2: SIM 200 mg+Ruxolitinib | Stage 2: SIM 700 mg+Ruxolitinib
Number analyzed (Participants) | 12 | 11 | 15 | 14
Percentage of participants
  Baseline : Screened Negative | 75.0 | 63.6 | 73.3 | 78.6
  Baseline : Screened Positive | 25.0 | 36.4 | 26.7 | 21.4
  Cycle 1 - Day 85 : Screened Negative: number analyzed (Participants) | 10 | 10 | 14 | 13
  Cycle 1 - Day 85 : Screened Negative | 100.0 | 90.0 | 57.1 | 92.3
  Cycle 1 - Day 85 : Screened Positive: number analyzed (Participants) | 10 | 10 | 14 | 13
  Cycle 1 - Day 85 : Screened Positive | 0 | 10.0 | 42.9 | 7.7
  Cycle 2 - Day 85 : Screened Negative: number analyzed (Participants) | 8 | 7 | 13 | 11
  Cycle 2 - Day 85 : Screened Negative | 100.0 | 85.7 | 69.2 | 90.9
  Cycle 2 - Day 85 : Screened Positive: number analyzed (Participants) | 8 | 7 | 13 | 11
  Cycle 2 - Day 85 : Screened Positive | 0 | 14.3 | 30.8 | 9.1
  Cycle 3 - Day 85 : Screened Negative: number analyzed (Participants) | 2 | 2 | 9 | 4
  Cycle 3 - Day 85 : Screened Negative | 100.0 | 100.0 | 100.0 | 75.0
  Cycle 3 - Day 85 : Screened Positive: number analyzed (Participants) | 2 | 2 | 9 | 4
  Cycle 3 - Day 85 : Screened Positive | 0 | 0 | 0 | 25.0
  Cycle 4 - Day 85 : Screened Negative: number analyzed (Participants) | 1 | 0 | 7 | 2
  Cycle 4 - Day 85 : Screened Negative | 100.0 |  | 100.0 | 100.0
  Cycle 4 - Day 85 : Screened Positive: number analyzed (Participants) | 1 | 0 | 7 | 2
  Cycle 4 - Day 85 : Screened Positive | 0 |  | 0 | 0
  Cycle 5 - Day 85 : Screened Negative: number analyzed (Participants) | 0 | 0 | 2 | 1
  Cycle 5 - Day 85 : Screened Negative |  |  | 100.0 | 100.0
  Cycle 5 - Day 85 : Screened Positive: number analyzed (Participants) | 0 | 0 | 2 | 1
  Cycle 5 - Day 85 : Screened Positive |  |  | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose date up to the last dose date (maximum: 94 weeks) plus 28 days
Description: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Arm/Group | Stage 1: SIM 200 mg | Stage 1: SIM 700 mg | Stage 2: SIM 200 mg+Ruxolitinib | Stage 2: SIM 700 mg+Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/12 | 1/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 8/12 | 1/12 | 5/15 | 4/15
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12 | 15/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: SIM 200 mg (N=12) | Stage 1: SIM 700 mg (N=12) | Stage 2: SIM 200 mg+Ruxolitinib (N=15) | Stage 2: SIM 700 mg+Ruxolitinib (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Periorbital infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: SIM 200 mg (N=12) | Stage 1: SIM 700 mg (N=12) | Stage 2: SIM 200 mg+Ruxolitinib (N=15) | Stage 2: SIM 700 mg+Ruxolitinib (N=15)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 5 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Systemic mastocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular hypokinesia (Cardiac disorders) | 1 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 2 | 4 | 5
Defaecation urgency (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 6 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 4 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 5 | 5 | 4
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 3 | 3
Asthenia (General disorders) | 1 | 1 | 4 | 0
Catheter site haematoma (General disorders) | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 2 | 0
Chills (General disorders) | 1 | 0 | 2 | 4
Cyst (General disorders) | 1 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 2 | 0
Fatigue (General disorders) | 5 | 3 | 5 | 8
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0
Infusion site pain (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 3 | 2 | 5 | 1
Pain (General disorders) | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 2 | 0 | 1
Pyrexia (General disorders) | 4 | 2 | 2 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 5 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0
Pneumonia cryptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 5 | 2
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 3 | 2
Urinary tract infection (Infections and infestations) | 4 | 0 | 4 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 3
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural oedema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 3 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram qt prolonged (Investigations) | 0 | 2 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 6 | 3 | 2 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 2
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 3 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2 | 2
Paraesthesia (Nervous system disorders) | 2 | 2 | 3 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
White matter lesion (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 2
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 3 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urethral disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 5 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 4 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 2 | 1
Hypertension (Vascular disorders) | 1 | 1 | 2 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1
Intra-abdominal haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Temporal arteritis (Vascular disorders) | 1 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years